CLINICAL TRIAL: NCT05725759
Title: The Effects of Rehabilitation on Functional Outcomes in Patients With SOD1 ALS Treated With Tofersen
Brief Title: Rehabilitation in SOD1 ALS Treated With Tofersen
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Sean E Smith, Instructor in Neurology, Washington University School of Medicine
Other Study IDs: 202208170
Record Dates: First submitted 2023-02-01; First posted 2023-02-13 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Amyotrophic Lateral Sclerosis; Lou Gehrig Disease; Familial Amyotrophic Lateral Sclerosis; Motor Neuron Disease; Motor Neuron Disease, Familial
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease | interventions — Rehabilitation; Physical Therapy Modalities; Occupational Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rehabilitation Arm: Participants will participate in outpatient physical and/or occupational therapies while participating in the tofersen early access program (EAP)
  Interventions: Behavioral: Rehabilitation

INTERVENTIONS:
Behavioral: Rehabilitation — Particapants currently receiving tofersen treatment will be referred to outpatient physical and/or occupational therapy.
  Other Names: physical therapy; occupational therapy

SUMMARY:
The primary objective of this study is to document and describe the effects of a personalized rehabilitation program for patients with SOD1 ALS participating in the tofersen expanded access program. Participants currently receiving tofersen treatment will be referred to outpatient physical and/or occupational therapy. Participants will have an initial assessment performed and an individualized rehabilitation program will be prescribed. Each participant is encouraged to follow the prescribed recommendations that will include scheduled outpatient therapy sessions, functional assessments, and/or a home-based rehabilitation program. Functional assessments will be done at a minimum of every three months.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of ALS with an SOD1 mutation
* Current enrollment in the tofersen expanded access program
* Age greater than 18 years
* Medically able to participate in outpatient physical therapy and/or home-based rehabilitation, as determined by the treating health care provider

Exclusion Criteria:

* Any comorbidities or conditions that, in the opinion of the treating healthcare provider, would unacceptably increase the risk of participation in outpatient physical therapy and/or home-based rehabilitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with SOD1 ALS
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2022-11-08 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Amyotrophic Lateral Sclerosis Functional Rating Scale - Revised (ALSFRS) | 12 months
  ALSFRS-R measures functional disease severity in four functional domains, bulbar function, gross motor skills, fine motor skills, and respiratory. The assessment contains 12 questions scored from 0 (no function) to 4 (full function), with a total possible score of 48, which will indicate the highest level of function.

SECONDARY OUTCOMES:
1. Change from baseline in Handheld Dynamometry (HHD) | 12 months
  Quantitative muscle strength will be evaluated using HHD of multiple muscles using standard participant positioning.
2. Change from baseline in Rasch-Built Overall Amyotrophic Lateral Sclerosis Functional Rating (ROADS) | 12 months
  ROADS measures disability across multiple daily activities. For each question, response options are as follows: 0=unable to perform; 1=abnormal, able to perform but with difficulty; and 2=normal, able to perform without difficulty.
3. Change from baseline in ALS Assessment Questionnaire, 5-item (ALSAQ-5) | 12 months
  Quality of life will be measured using the 5-item Amyotrophic Lateral Sclerosis Assessment Questionnaire (ALSAQ-5) patient-reported outcome (PRO)
Change from baseline in motor Functional Independence Measure (motor FIM) | 12 months
  Measures level of disability and indicates level of assistance required to perform activities of daily living.
Change from baseline in Modified Ashworth Scale (MAS) | 12 months
  The MAS is 6-point scale that that grades spasticity, scored from 0 to 4, where 0 is normal muscle tone and 4 is severe increase in muscle tone
Change from baseline in Slow Vital Capacity (SVC) | 12 months
Change from baseline in Maximal Inspiratory Pressure (MIP) | 12 months
Change from baseline in Fatigue Severity Scale (FSS) | 12 months
  FSS measures how fatigue interferes with activities. It is a 9-item questionnaire scored on a 7-point scale, 1 = strongly disagree to 7 = strongly agree, and the higher the score equal to the greater the severity of fatigue

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- See also: Washington University ALS Center website — https://alscenter.wustl.edu